CLINICAL TRIAL: NCT00794105
Title: Observation of Gas Exchange in the Middle Ear
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: David Cohen, MD, Shaare Zedek Medical Center
Other Study IDs: cohenmed.CTIL
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Normal Middle Ears.; Otitis Media Ears.
Keywords: Gas; Middle ear
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal ears
- Otitis media ears.

SUMMARY:
Observation of fluid behavior over a perforated eardrum.

A comparison of the behavior of the gas in normal vs. different kinds of otitis media ears.

DETAILED DESCRIPTION:
Fluid present in middle ears is observed during the regular treatment of patients.

The observation in made during the treatment and not as an additional activity. The fluid is either a steroids solution or sterile normal saline or ear's mucus discharge, all in perforated eardrums, either as a part of their intra-tympanic treatment for sudden hearing loss, or traumatic perforation [considered as the normal ears] compared to otitis media ears.

The observation is made on bubble formation over the perforation. The time length of the inspection is about 1 minute, under the microscope, during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients having perforated eardrum.

Exclusion Criteria:

* Non cooperative patients.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated as a routine treatment in the outpatient or patients admitted for treatment of sudden hearing loss.
Sampling Method: Non-Probability Sample
Dates: Start 2008-11

PRIMARY OUTCOMES:
Creation of air bubbles. | one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Otolaryngology Dept., Shaare Zedek Medical Center, Jerusalem, Israel